CLINICAL TRIAL: NCT05689944
Title: Effect of Dance-therapy on Chronic Adolescent Pain Patients - a Randomized Controlled Trial Study
Brief Title: Dance-therapy and Chronic Pain
Acronym: ALGODANCE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 69HCL22_0361
Record Dates: First submitted 2022-12-01; First posted 2023-01-19 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Chronic Pain; Complex Regional Pain Syndromes; Tension-Type Headache
Keywords: Dance-therapy; Chronic pain; Complex Regional Pain Syndrome; Tension Type Headache; Adolescents
MeSH Terms: conditions — Chronic Pain; Complex Regional Pain Syndromes; Tension-Type Headache | interventions — Dance Therapy; Art Therapy; Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): Patients in the control group will not participate in any art-therapy or yoga interventions. They will be asked to complete pain and sleep diaries, questionnaires and pain, fatigue and mood scales at the same times and for the same duration as the other groups.
- Dance-therapy group (Experimental): Patients in the dance-therapy group will attend a weekly session of dance-therapy between weeks 1 and 15 of the protocol (15 sessions). They will be asked to complete daily pain and sleep diaries at weeks W0, W5, W16, W20 and W28 as well as questionnaires (kinesiophobia, anxiety, catastrophizing, fear of pain, quality of life, body image/self-perception). They will also be asked to assess their pain, fatigue and mood levels at the end of each week between W1 and W15.
  Interventions: Behavioral: Dance-therapy
- Art-therapy group (Experimental): Patients in the art-therapy group will attend a weekly session of art-therapy (drawings, collages…) between weeks 1 and 15 of the protocol (15 sessions). They will be asked to complete daily pain and sleep diaries at weeks W0, W5, W16, W20 and W28 as well as questionnaires (kinesiophobia, anxiety, catastrophizing, fear of pain, quality of life, body image/self-perception). They will also be asked to assess their pain, fatigue and mood levels at the end of each week between W1 and W15.
  Interventions: Behavioral: Art-therapy
- Yoga group (Experimental): Patients in the yoga group will attend a weekly session of Vinyasa yoga between weeks 1 and 15 of the protocol (15 sessions). They will be asked to complete daily pain and sleep diaries at weeks W0, W5, W16, W20 and W28 as well as questionnaires (kinesiophobia, anxiety, catastrophizing, fear of pain, quality of life, body image/self-perception). They will also be asked to assess their pain, fatigue and mood levels at the end of each week between W1 and W15.
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Dance-therapy — This session will take place once a week between weeks 1 and 15 of the protocol.
  * 5 mn of welcome and presentation of the upcoming session
  * 5 mn of self-evaluation of the pain as well as of the thymia and the fatigue before the beginning of the session (Visual numerical scales: VNS)
  * 15 mn of body warm-up with taught contemporary dance exercises
  * 15 mn of creative research based on dance improvisation on a given theme
  * 15 mn of sharing for the elaboration of a choreography
  * At the end of the session, 5mn of self-evaluation of the pain, the thymia, the fatigue and the level of appreciation of the session (VNS).
  After the session, the patient will be asked to think about the next session if he/she wishes (e.g. think of a choreography, remember what was done etc. ....) in order to encourage the commitment to care. These sessions will be based on contemporary dance and dance improvisation techniques.
  Arms: Dance-therapy group
Behavioral: Art-therapy — This session will take place once a week between weeks 1 and 15 of the protocol.
  * 5 mn of welcome and presentation of the upcoming session
  * 5 mn of self-evaluation of the pain as well as of the thymia and the fatigue before the beginning of the session (Visual numerical scales: VNS)
  * 10 mn of discovery of a new technique (acrylic painting or collage).
  * 35 mn of practice in a project fixed beforehand
  * At the end of the session, 5mn of self-evaluation of the pain, the thymia, the fatigue and the level of appreciation of the session (VNS).
  After the session, the patient will be asked to think about the next session (e.g. collecting plants for collage....) in order to encourage commitment to the treatment. The sessions will be based on acrylic painting or collage techniques.
  Arms: Art-therapy group
Behavioral: Yoga — This session will take place once a week between weeks 1 and 15 of the protocol.
  * 5 mn welcome
  * 5 mn of self-evaluation of the pain as well as of the thymia and the fatigue before the beginning of the session (Visual numerical scales: VNS)
  * 50 mn of Vinyasa type yoga (warm-up, breathing, balance, strength and flexibility, relaxation)
  * 5 mn of closing of the session
  * At the end of the session, 5mn of self-evaluation of the pain thanks, the thymia, the fatigue and the level of appreciation of the session (VNS).
  These sessions engage the body without entering into a therapy protocol turned towards art as in the two previous interventions.
  Arms: Yoga group

SUMMARY:
Pain, when it becomes chronic, can be a threat to patients and it is very common to observe a fear of pain and a fear of movement (kinesiophobia). Avoidance of movement due to fear of pain can lead to a deterioration of body image. Non-medicinal therapies are essential to correct this fear and movement avoidance behavior, to decrease "catastrophic" judgments and thus anxiety. The use of art-therapy in the accompaniment of patients with pain has shown, in particular, decreases in the intensity of pain, the level of anxiety, an improvement in stress, mood and overall psychological state. However, according to the current literature, it appears that 1) this technique is rarely used in children or adolescents, for whom non-medicinal therapies are fundamental, and 2) in the case of chronic pain, the form of art used is very rarely related to the body (most often painting, drawing, music...).

In this project, investigators propose to set up and test the potential benefit of art-therapy sessions related to the body, namely dance-therapy, in adolescents and young adults suffering from chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12 to 20 years, girls or boys, with either complex regional pain syndrome (CRPS) or chronic tension-type headache (CTTH).
* Diagnosis of CRPS or chronic CTTH made in a Pain Management Center
* Patients followed in a Pain Management Center (to ensure that patients entering the protocol have pain that is not relieved by conventional treatments)
* Patients who have given written consent for adults or whose parents have given consent for minors
* Patients who are affiliated with or benefit from a social security system.

Exclusion Criteria:

* Patients with headaches other than CTTH
* Patients with other neurological or psychological disorders
* Patients with psychiatric illnesses
* Patients with chronic pain conditions other than CRPS or CTTH
* Patients with chronic infectious, metabolic, cancerous, autoimmune diseases.
* Patients whose motor limitations are not related to the diagnosis of CRPS or CTTH (e.g. cerebral palsy, spinal cord injury...)
* Non-communicating patients including deaf and hard of hearing patients
* Patients or parents who do not speak or read French
* Pregnant women
* Dance or yoga professionals (dance or yoga teachers or those studying to become teachers)

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Assesment of pain change | Weeks 0, 5, 16, 20 and 28.
  Daily self-assessment on visual numerical scale of pain intensity upon awakening, at bedtime, and on average during the day. Each item is scored 0-10 (0= no pain; 10 = maximal pain). Reporting of the times during the day and night when the patient feels pain and its intensity.

SECONDARY OUTCOMES:
Kinesiophobia | Inclusion, weeks 5, 16, 20, 28.
  Evaluation of the kinesiophobia index with the TAMPA scale: 13 items to be evaluated on a 4-point Likert-type scale between 1 (strongly disagree) and 4 (strongly agree). Scores between 13 and 52, a score of 30/52 being considered as a significant kinesiophobia.
Anxiety (adolescents) | Inclusion, weeks 5, 16, 20, 28
  Screen for Child Anxiety Related Disorders (SCARED). 41 items to be evaluated on a 3-point Likert-type scale between 0 ('not true' or 'almost never true') and 2 ('very true' or 'often true'). A score greater than or equal to 25 may indicate the presence of an anxiety disorder.
Anxiety (adults) | Inclusion, weeks 5, 16, 20, 28
  For adult patients: HAD scale. 14 items rated from 0 to 3. Seven items relate to anxiety and seven others to the depressive dimension. The highest scores correspond to the presence of a more severe symptomatology.
Pain catastrophizing | Inclusion, weeks 5, 16, 20, 28.
  Pain catastrophizing scale (PCS). 13 items to be evaluated on a 5-point Likert-type scale between 0 (never) to 4 (always). Scores between 0 and 52. A total PCS score of 30 represents clinically relevant level of catastrophizing.
Fear of Pain (adolescents) | Inclusion, weeks 5, 16, 20, 28.
  Fear of Pain Questionnaire (FOPQ). 24 items to be evaluated on a 5-point Likert-type scale between 0 (Strongly disagree) and 4 (Strongly agree). Scores between 24 and 96. A total score between 51 and 96 represents a high fear of pain
Fear of Pain (adults) | Inclusion, weeks 5, 16, 20, 28.
  For adults patients: FABQ questionnaire. 16 items evaluated on a 7-point Likert scale between 0 (strongly disagree) and 4 (strongly agree). The first 5 items test fear and beliefs about pain in relation to physical activity and the second part of the questionnaire (12 items) tests fear and beliefs about pain in relation to work.
Incidence of art therapy on quality of life (adolescents) | Inclusion, weeks 5, 16, 20, 28.
  -VSP-A scale for adolescents. 40 items to be evaluated on a 5-point Likert-type scale between 0 (always) and 100 (never). This scale explores 6 areas (psychological well-being, energy/vitality, leisure activities, friendships, relationships with parents, school life). The scores are averaged and then transformed to obtain a rating between 0% and 100%. A total score below 50% is considered to reflect a low quality of life.
Incidence of art therapy on quality of life (adults) | Inclusion, weeks 5, 16, 20, 28.
  -The McGill Quality of Life Questionnaire-revised version (MQOL-R) for the adults. 14 items to be evaluated on a 11-point Likert-type scale between 0 (not at all) and 10 (extremely). These items form 4 subscales (physical, psychological, existential, and social). The total MQOL-R score is the average of the scores on the 4 subscales.
Body satisfaction and global self-perception | Inclusion, weeks 5, 16, 20, 28.
  QSCPGS questionnaire. 20 items. The QSCPGS is divided into two parts. Each part consists of a series of 10 items. The first set is designed to define how the individual perceives his or her body and the second seeks to highlight the feelings of himself in a more global way. Each item is composed of a positive term (good health, pure, calm. . .) and its opposite (bad health, impure, nervous. . .); these two expressions are opposed by a series of numbers from 1 to 5 presented in mirror and separated in their center by the 0; the 1 corresponds to the answer "very little" and 5: "very strong".
Incidence of art therapy on sleep quality | Weeks 0, 5, 16, 20 and 28.
  Daily measurement of sleep quality, wake quality and average day energy (5-point Likert-type scale between 'very good' and 'very bad'). Filling out a sleep diary with the daily bedtime and wake-up times for one week.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuroscience Research Center of Lyon (CRNL)- INSERM U1028 - NEUROPAIN laboratory, Bron, France

IPD SHARING:
Plan to Share IPD: No